CLINICAL TRIAL: NCT05290558
Title: The Therapeutic Effects of Bu Shen Yi Jing Pill on Semen Quality in Sub Fertile Males: a Randomized Controlled Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/2019
Record Dates: First submitted 2021-12-29; First posted 2022-03-22 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Male Infertility; Infertility; Traditional Chinese Medication (TCM); Reproductive Issues
Keywords: Infertility; Sperm; Traditional Medicine
MeSH Terms: conditions — Infertility, Male; Infertility | interventions — Drug and Narcotic Control

STUDY DESIGN:
Intervention Model Description: This is a double-blinded randomised control trial. Participants will be randomised using block randomization by a pre-determined randomisation schedule generated by a biostatistician in block size of 4. Enrolment and assignment of intervention will be carried out by an investigator. The investigators will perform block randomization of the subjects in blocks of 4 in the ratio of 1:1 such that 2 will be assigned to treatment and 2 will be assigned to placebo.
Who Masked: Participant, Care Provider
Masking Description: This is a double-blind study. The randomization master list will be kept with the investigator and both patients and physician will be blinded to the treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients in this arm will be given a placebo pill that resembles the actual Bu Shen Yi Jing Pill.
  Interventions: Drug: Placebo Drug
- Bu Shen Yi Jing Pill (Active Comparator): Patients in this arm will be given the BSYJ Pill.
  Interventions: Drug: Bu Shen Yi Jing Pill

INTERVENTIONS:
Drug: Bu Shen Yi Jing Pill — Bu Shen Yi Jing Pill contained Radix Pseudostellaria, Fructus Lycii, Radix Et Rhizoma Salviae, Rhizoma Dioscorea, Semen Plantaginis, Semen Cuscuta, Patriniae Herba, Herba Epimedii, Radix Ophiopogonis, Fructus Rubi, Fructus Corni, Bupleurum roots, Fructus Schisandrae Chinensis, Radix Et Rhizoma Glycyrrhizae.
  Dosage of the study drug is as follows: 3 pills each time, for 3 times a day, taken for 6 days every week for 1 year
  Other Names: BSYJ Pill
  Arms: Bu Shen Yi Jing Pill
Drug: Placebo Drug — Placebo contains the ingredients: grounded black rice and permitted colouring. The ingredients are encapsulated within a gelatine capsule.
  Dosage of the study drug is as follows: 3 pills each time, for 3 times a day, taken for 6 days every week for 1 year
  Other Names: Control drug
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety and efficacy of Bu Shen Yi Jing (BSYJ) Pill , a type of traditional Chinese medicine, in improving male subfertility and semen parameters.

DETAILED DESCRIPTION:
Subfertility is defined as a failure to conceive after 1 year of regular unprotected intercourse. Impaired fertility affects 10 to 15% of couples and male factor is the cause of subfertility in 25 to 40% of couples. With increasing paternal age, semen volume, sperm motility and the percentage of sperm with normal morphology decreases. The majority of men who present with subfertility have either abnormal sperm density, motility or morphology, or a combination of the above, and treatment for this condition is varied and empirical.

There is a paucity of studies and randomized controlled trials to guide treatment of male factor subfertility. Various antioxidant formulations and multivitamins have been used empirically but have not been shown consistently to improve sperm counts and viability. When treatment fails, assisted reproduction will be the last resort. All assisted reproduction treatments are associated with medical, financial and emotional burden. Given the lack of proven treatment options in Western Medicine, Traditional Chinese Medicine (TCM) may provide a viable complementary treatment option. One such option is the Bu Shen Yi Jing (BSYJ) pill.

A clinical observational study conducted by the team in Singapore Thong Chai Medical on subfertile male patients with poor sperm quality and a body constitution of Kidney Deficiency showed that 2 courses of BSYJ pill over a 6 months' duration resulted in successful conception of 33% of azoospermic male patients (n = 60). In a subgroup of patients where serial sperm analysis was available (n=10), the percentage of sperm with grade A motility increased from a median of 22.6 ± 2.4% pre-treatment to 35.1 ± 3.2% post treatment (p < 0.05); and the hyaluronic binding assay improved from 33.2 ± 2.4% to 72 ± 4.6% (p < 0.05). This suggests that BSYJ pills possibly works on improving the motility of the sperms in patients having the Kidney deficiency body constitution.

As such, this study aims to validate these hypotheses and anecdotal evidence by conducting a safety and efficacy study of the BSYJ pill on a prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Duration of subfertility (both primary and secondary) ≥ 1 year;
* Any or combination of the three abnormal semen parameters, defined according to the 2010 WHO criteria, including

  * Oligozoospermia, with sperm concentration less than 15 x 10^6,
  * Teratozoospermia, with normal sperm morphology less than 4%, and
  * Asthenozoospermia, with total sperm motility less than 40%, or progressive sperm motility less than 32%.
* Diagnosed with TCM syndrome of Kidney Deficiency Based on a prominent TCM diagnosis textbook known as TCM Diagnostics, the main symptoms patients need to fulfil for Kidney Deficiency are either nocturnal polyuria or lower back pain. In addition, patients need to fulfil any 1 of the secondary symptoms, including fatigue; dizziness; tinnitus or deafness; memory loss; excessive urination; low libido; wet dreams; premature ejaculation; presence of feverish palms and soles or night sweats; dry mouth or throat; cold intolerance or preference for warmth; poor sleep quality. Presence of both 1 main symptom and 1 secondary symptom allows for the diagnosis of the Kidney Deficiency syndrome.

Patients who meet all three criteria mentioned above will be included in the study.

Exclusion Criteria:

* Azoospermia and severe oligoasthenoteratozoospermia;
* Aspermia;
* Varicocele;
* Recent urogenital infections;
* Y chromosome deletions;
* Abnormal karyotypes
* History of chemotherapy and / or radiotherapy;
* Patients on fertility supplements or supplements marketed to improve fertility;
* Patients with uncontrolled diabetes or/and hypertension; with uncontrolled chronic medical conditions
* Patients currently already on BSYJ pills treatment

Ages: 21 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the change in sperm volume from baseline after treatment with BSYJ pill | 1 year
  From sperm samples analyses
To determine the change in sperm morphology from baseline after treatment with BSYJ pill | 1 year
  From sperm samples analyses
To determine the change in sperm motility from the baseline after treatment with BSYJ pill | 1 year
  From sperm samples analyses
To determine the change in sperm concentration from the baseline after treatment with BSYJ pill | 1 year
  From sperm samples analyses

SECONDARY OUTCOMES:
To determine the clinical pregnancy rate and successful delivery rate after BSYJ pill | 2 year
  Defined by the number of pregnancies and subsequent actual births after commencement of BSYJ pill
To study the safety and determine the changes in blood profile after treatment with BSYJ pill | 1 year
  Defined by changes in participant's full blood count, renal panel, liver function test and hormone profile.

OTHER OUTCOMES:
To assess the common side effects of the BSYJ pill | 1 year
  Participant reported symptoms of excessive heat syndrome such as ulcers and mouth dryness.
To assess the common gastrointestinal side effects of the BSYJ pill | 1 year
  Participant reported symptoms of gastrointestinal symptoms such as indigestion and appetite reduction.
To evaluate safety profile of BSYJ pill | Up to 1 year after recruitment
  Participants will be assessed frequently to pick up any side effects noted after commencement of BSYJ pill
Change from baseline severity based on TCM symptom scoring questionnaire | 1 year
  As BSYJ pills target the TCM syndrome of Kidney Qi deficiency, symptoms related to Kidney Qi deficiency syndrome, which includes frequent urination and back pain, fatigue and dizziness, may be improved through this research.
Number of participants with improvement in TCM syndrome of Kidney Qi deficiency from baseline according to the TCM symptom scoring questionnaire Stagnation | 1 year
  As BSYJ pills target the TCM syndrome of Kidney Qi deficiency, symptoms related to Kidney Qi deficiency syndrome, which includes frequent urination and back pain, fatigue and dizziness, may be improved through this research.
Patient's basic demographics | 1 year
  Defined by age, ethnicity, marital status
Patient's partner's basic demographics | 1 year
  Defined by age, ethnicity, marital status
Patients's anthropometry | 1 year
  Defined by height, weight and body mass index based on weight (kg) /height (m)2
Number of participants who smoke | 1 year
  Self-reported
Number of participants who take alcohol regularly | 1 year
  Self-reported based on the amount and frequency of alcohol intake
Number of participants who have dietary restrictions | 1 year
  Self-reported
Number of participants with occupational exposures to chemicals | 1 year
  Self-reported
Number of participants with exposure to hot baths or jacuzzi | 1 year
  Self-reported
Number of participants who uses recreational drugs | 1 year
  Self-reported
Number of participants who exercise regularly | 1 year
  Self-reported
Number of patients with significant medical history | 1 year
  Self-reported details of medical history
Number of patients with significant surgical history | 1 year
  Self-reported details of surgical history
Number of patients on regular medications | 1 year
  Self-reported details of types of regular medications
Number of patients with drug allergies | 1 year
  Self-reported details of drug allergies
Number of patients who take supplements | 1 year
  Self-reported details of the type of supplements taken
Number of patients who take steroids | 1 year
  Self-reported
Number of patients with previous history of sexually transmitted disease | 1 year
  Self-reported details of sexually transmitted disease
Number of patients with previous history of genital trauma | Since birth
  Self-reported details of genital trauma
Patient's fertility history | 1 year
  Determined by the number of years of attempts at conception, sexual intercourse frequency, number of paternity (including current and/or previous partners), previous fertility treatments and medications
Patient's partner's fertility history | 1 year
  Determined by the number of years of attempts at conception, sexual intercourse frequency, number of maternity (including current and/or previous partners), previous fertility treatments and medications, and menstrual history

CONTACTS AND LOCATIONS:
Overall Officials: Tat Xin Ee, MD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No